CLINICAL TRIAL: NCT01259687
Title: Pulse Transit Time in Anesthetized Ventilated Patients: Affect of Blood Pressure or Cardiac Output as Measured With NICOM Monitor
Brief Title: Pulse Transit Time in Anesthetized Patients: Blood Pressure or Cardiac Output as Measured With NICOM Monitor
Acronym: PuTT-NICOM
Status: Completed | Type: Observational
Sponsor: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Pizov Reuven, MD, Clinical Professor of Anesthesiology, Carmel Medical Center
Other Study IDs: CMC-09-0124-CTIL
Record Dates: First submitted 2010-12-07; First posted 2010-12-14 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2013-11

CONDITIONS: Anesthetized Ventilated Patients
Keywords: Electrocardiogram; Arterial line waveform; Cardiac output

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study group
  Interventions: Device: Non-invasive cardiac output monitoring

INTERVENTIONS:
Device: Non-invasive cardiac output monitoring — During the surgery the continuous monitoring of blood pressure by peripheral artery catheter and cardiac output by NICOM (non-invasive cardiac output monitoring) will be applied. In case of intraoperative hemodynamic changes (hypertension, hypotension) the patient will be treated according to the standard care by Phenylephrine, Nitroglycerine or Colloid fluid boluses. Cardiac output will be measured by NICOM just before and after each treatment of hemodynamic events that described above. Simultaneous records of ECG, arterial and plethysmographic waveforms will be made just before and after each event. Systolic blood pressure and PuTT will be measured OFFLINE from the recorded waveforms
  Other Names: Cheetah Reliant; NICOM; Cheetah Medical

SUMMARY:
Pulse transit time (PuTT) - the time between R wave on ECG and initiation of upstroke in the peripheral arterial waveform - described in the previous studies as value that reflects changes in both blood pressure and blood volume. The investigators are assuming that PuTT changes reflect the dynamic of systolic blood pressure but not cardiac output fluctuations.

DETAILED DESCRIPTION:
Background Pulse transit time (PuTT) - the time between R wave on ECG and initiation of upstroke in the peripheral arterial waveform - described in the previous studies as value that reflects changes in both blood pressure and blood volume. We are assuming that PuTT changes reflect the dynamic of systolic blood pressure but not cardiac output fluctuations.

Clinical trial objectives Investigate a link between PuTT (Pulse transit time) and changes in blood pressure and cardiac output measured by non-invasive cardiac output monitoring device (NICOM).

Endpoints PuTT Blood pressure: systolic, diastolic, mean Heart rate Cardiac output-Index Systemic vascular resistance-Index

Prospective nonrandomized clinical trial

Inclusion criteria Need for continuous invasive monitoring of blood pressure - according to the type of surgery the patient's health status Normal sinus rhythm

Exclusion criteria Pregnancy Cave to Nitroglycerine or Phenylephrine Chronic renal failure with creatinine level above 2 mg%

Safety assessment methods Monitoring of cardiac output is one of the most important elements of hemodynamic monitoring. In the past this monitoring was based mainly on the invasive and awkward methods causing usage only in exceptional cases. NICOM device allows accurate non-invasive monitoring of cardiac output During anesthesia patient care changes are made according to changes in vital indicators such as blood pressure, pulse, cardiac output. So during the study, anesthesia care can be affected by the indices obtained using a NICOM.

Data processing and analysis During the surgery the continuous monitoring of blood pressure by peripheral artery catheter and cardiac output by NICOM will be applied.

In case of hemodynamic changes the patient will be treated according to the standard care:

In case of decrease of systolic blood pressure below 80 mmHg (in the patients with history of arterial hypertension - below 90 mmHg) and HR is above 70 bpm the patient will be treated by repeated boluses of Phenylephrine 50-100 mcg until the systolic blood pressure will increase by at least 20%.

Intraoperative hypertension above 160 mmHg will be treated by repeated boluses of Nitroglycerine 100 mcg until the systolic blood pressure will decrease by at least 20%.

Hypovolemia will be treated by boluses of colloid solution - HAES 6% - at dose of 7 ml/kg of body mass during 15 min.

Study procedures

Cardiac output will be measured by NICOM just before and after each treatment of hemodynamic events that described above. Simultaneous records of ECG, arterial and plethysmographic waveforms will be made just before and after each event.

Systolic blood pressure and PuTT will be measured OFFLINE from the recorded waveforms.

ELIGIBILITY:
Inclusion Criteria:

* All patients scheduled for elective surgery and require invasive monitoring of blood pressure according to their medical condition and type of surgery

Exclusion Criteria:

* Patients under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing various types elective surgery which require continous invasive monitoring of blod pressure
Sampling Method: Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2011-01; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Pulse transit time (PuTT) | Two minutes after each intervention (giving Nitroglycerine, Phenylephrine or Fluid loading)
  Simultaneous record of arterial line waveform and ECG will be made just before and 2 minute after giving one of treatments (Phenylephrine, Nitroglycerine or fluid bolus). PuTT will be measured offline from the record

CONTACTS AND LOCATIONS:
Overall Officials: Reuven Pizov, MD, Principal Investigator — Carmel Medical Center
Locations (2):
- Israel (2):
  - Carmel Medical Center, Haifa
  - The Lady Davis Carmel Medical Center, Haifa